CLINICAL TRIAL: NCT01454869
Title: Efficacy of Heparin Nebulization on Lung Injury Score in Inhalation Burn Injury
Brief Title: The Effect of Heparin on Inhalation Injury
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to insufficient funds
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 89-04-129-12415
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Heparin
Keywords: heparin
MeSH Terms: interventions — Standard of Care; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): nac + salotamul
  Interventions: Drug: standard care
- heparin group (Experimental): heparin group
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: standard care — Standard care treatment consist of chest physiotherapy ,early ambulation, airway suctioning, bronchial hygiene therapy , salbutamol nebulization(100-200 µgQ4h)/N-acetyl cysteine20% nebulization(3cc Q4h) and if needed mechanical ventilation support.
  Other Names: routin
  Arms: Standard care
Drug: Heparin — Study group would consist of 85 burn patients with documented smoke inhalation injury who will be randomized to receive standard care plus heparin nebulization(5000U every 4 hours for 7 days) in combination with intravenously administrated fresh frozen plasma(10 cc/Kg daily for 7 days).
  Other Names: new
  Arms: heparin group

SUMMARY:
This is a prospective randomized clinical trial about the efficacy of heparin nebulization on lung injury score in inhalation burn injury in Mothary burn hospital. This study would consist of 170 burn patients with documented inhalation injury in 2 arms (control group and study group). Allocation ratio is1:1. Masking was not possible. The patients' primary outcome will be assessed for Lung Injury Scale and the patients' secondary outcome will be assessed for mortality, Coagulation tests (PT, PTT), ICU and hospital stay and duration of mechanical ventilation support. Duration of this study is about 32 months.

DETAILED DESCRIPTION:
This study would consist of 170 burn patients with documented smoke inhalation injury who will be randomized to receive either standard care alone (control group) or standard care plus heparin nebulization in combination with intravenously administrated fresh frozen plasma (study group). Standard care treatment consist of: chest physiotherapy ,early ambulation, airway suctioning, bronchial hygiene therapy , salbutamol nebulization (100-200 µgQ4h)/N-acetyl cysteine 20% nebulization (3cc Q4h) and if needed mechanical ventilation support. Study care treatment consist of: Standard care + Heparin nebulized administration(5000U every 4 hours for 7 days) and fresh frozen plasma intravenously administration (10 cc/Kg daily for 7 days) The patients' primary outcome will be assessed for Lung Injury Scale (LIS) every day by using fallowing parameters: (1) chest X-ray evaluated for alveolar consolidation (2) ratio of the partial pressure of oxygen in arterial blood to the inspiratory fraction of oxygen (3) PEEP level if ventilated (4) respiratory compliance if known Parameter Finding Value Rx.Torax no alveolar consolidation 0 alveolar consolidation de 1 quadrant 1 alveolar consolidation de 2 quadrant 2 alveolar consolidation de 3 quadrant 3 alveolar consolidation de 4 quadrant 4 Hypoxemia PaO2/FIO2 > 300 0 PaO2/FIO2 225 - 299 1 PaO2/FIO2 175 - 224 2 PaO2/FIO2 100 - 174 3 PaO2/FIO2 < 100 4 PEEP PEEP <= 5 cm H2O 0 PEEP 6 - 8 cm H2O 1 PEEP 9 - 11 cm H2O 2 PEEP 12 - 14 cm H2O 3 PEEP >= 15 cm H2O 4 Compliance >= 80 mL/cm H2O 0 compliance 60 - 79 mL/cm H2O 1 compliance 40 - 59 mL/cm H2O 2 compliance 20 - 39 mL/cm H2O 3 compliance <= 19 mL/cm H2O 4 2 The patients' secondary outcome will be assessed for mortality(for 28 days post injury), Coagulation tests(PT,PTT) (for 7 days post injury),ICU and hospital stay(for 7 days post injury) and duration of mechanical ventilation support(for 7 days post injury). In each group 85 Patients will be selected by simple randomization. Allocation ratio is1:1. Blinding of this study was not possible.

PEEP: positive end expiratory pressure- PaO2: partial pressure of oxygen in arterial blood- FIO2: inspiratory fraction of oxygen PT: prothrombin time- PTT: partial thrombin time- ICU: intensive care unite- Rx: X-Ray

ELIGIBILITY:
Inclusion Criteria:

* Burn patients admitted to Motahary burn center with documented inhalation injury (as defined by clinical or bronchoscopic evaluation)

Exclusion Criteria:

* Non-survivable burn patients;
* history of coagulation disease;
* chronic obstructive pulmonary disease(COPD);
* pneumonia diagnosed at admission;
* inability to confirm definitive diagnosis of inhalation injury and co poisoning or Cyanide hydrogen intoxication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Lung Injury Score | Daily untill 7 days post injury
  (1) chest X-ray evaluated for alveolar consolidation (2) ratio of the partial pressure of oxygen in arterial blood to the inspiratory fraction of oxygen (3) PEEP level if ventilated (4) respiratory compliance

SECONDARY OUTCOMES:
Mortality | 28 days post injury
  Physical exam & EKG
pt/ptt | Up to 7 days post injury
  Daily
Duration of mechanical ventilation | 7 days post injury
Duration of hospital stay | 7 days post injury

CONTACTS AND LOCATIONS:
Overall Officials: Seyed H Salehi, MD, Study Chair — Burn research of Tehran university of Medical Sciences
Locations (1):
- Shahid Mothary Burn Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Maybauer MO, Rehberg S, Traber DL, Herndon DN, Maybauer DM. [Pathophysiology of acute lung injury in severe burn and smoke inhalation injury]. Anaesthesist. 2009 Aug;58(8):805-12. doi: 10.1007/s00101-009-1560-x. German. PMID 19517070
- [Background] Brown M, Desai M, Traber LD, Herndon DN, Traber DL. Dimethylsulfoxide with heparin in the treatment of smoke inhalation injury. J Burn Care Rehabil. 1988 Jan-Feb;9(1):22-5. doi: 10.1097/00004630-198801000-00007. PMID 3356738
- [Background] Enkhbaatar P, Esechie A, Wang J, Cox RA, Nakano Y, Hamahata A, Lange M, Traber LD, Prough DS, Herndon DN, Traber DL. Combined anticoagulants ameliorate acute lung injury in sheep after burn and smoke inhalation. Clin Sci (Lond). 2008 Feb;114(4):321-9. doi: 10.1042/CS20070254. PMID 17927568
- [Background] Desai MH, Mlcak R, Richardson J, Nichols R, Herndon DN. Reduction in mortality in pediatric patients with inhalation injury with aerosolized heparin/N-acetylcystine [correction of acetylcystine] therapy. J Burn Care Rehabil. 1998 May-Jun;19(3):210-2. doi: 10.1097/00004630-199805000-00004. PMID 9622463
- [Background] Cancio LC. Airway management and smoke inhalation injury in the burn patient. Clin Plast Surg. 2009 Oct;36(4):555-67. doi: 10.1016/j.cps.2009.05.013. PMID 19793551
- [Background] Toon MH, Maybauer MO, Greenwood JE, Maybauer DM, Fraser JF. Management of acute smoke inhalation injury. Crit Care Resusc. 2010 Mar;12(1):53-61. PMID 20196715
- [Background] Muller MJ, Pegg SP, Rule MR. Determinants of death following burn injury. Br J Surg. 2001 Apr;88(4):583-7. doi: 10.1046/j.1365-2168.2001.01726.x. PMID 11298629
- [Background] Tredget EE, Shankowsky HA, Taerum TV, Moysa GL, Alton JD. The role of inhalation injury in burn trauma. A Canadian experience. Ann Surg. 1990 Dec;212(6):720-7. doi: 10.1097/00000658-199012000-00011. PMID 2256764
- [Background] Shirani KZ, Pruitt BA Jr, Mason AD Jr. The influence of inhalation injury and pneumonia on burn mortality. Ann Surg. 1987 Jan;205(1):82-7. doi: 10.1097/00000658-198701000-00015. PMID 3800465
- [Background] Darling GE, Keresteci MA, Ibanez D, Pugash RA, Peters WJ, Neligan PC. Pulmonary complications in inhalation injuries with associated cutaneous burn. J Trauma. 1996 Jan;40(1):83-9. doi: 10.1097/00005373-199601000-00016. PMID 8577005
- [Background] Murakami K, Enkhbaatar P, Shimoda K, Mizutani A, Cox RA, Schmalstieg FC, Jodoin JM, Hawkins HK, Traber LD, Traber DL. High-dose heparin fails to improve acute lung injury following smoke inhalation in sheep. Clin Sci (Lond). 2003 Apr;104(4):349-56. PMID 12653676
- [Background] Janne O, Kontula K, Vihko R. Review article: mechanism of action of female sex steroids. Acta Obstet Gynecol Scand Suppl. 1976;51:29-45. No abstract available. PMID 180744